CLINICAL TRIAL: NCT04045340
Title: Intraoperative Transesophageal Echocardiography in On-pump Mitral Surgery: A Single Center Prospective Observational Study of Global Longitudinal Strain and Global Longitudinal Strain Rate as Predictors of Unfavorable Outcome
Brief Title: Intraoperative Global Longitudinal Strain and Global Longitudinal Strain Rate as Predictors of Unfavorable Outcome in On-Pump Mitral Surgery
Acronym: Mit-GO
Status: Completed | Type: Observational
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Fabrizio Monaco, Head of Cardiac and Vascular Anestesia, Scientific Institute San Raffaele
Other Study IDs: MIT-GO-2019
Record Dates: First submitted 2019-07-26; First posted 2019-08-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2020-10

CONDITIONS: Mitral Valve Disease; Low Cardiac Output Syndrome
MeSH Terms: conditions — Cardiac Output, Low | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Device: Philips QLAB Ultrasound Quantification Software — Offline processing of intraoperative transesophageal echocardiography would be performed with Global Longitudinal Strain on apical 4 chamber, apical 2 chamber and long axis views in order to analyze left ventricle and left atrium contractility and right ventricle free wall motion
  Other Names: Echocardiography

SUMMARY:
The aim of the present study is to assess the best echocardiographic parameters (GLS, GLS rate and standard echocardiographic parameters) predicting LCOS in on-pump mitral surgery.

DETAILED DESCRIPTION:
Low cardiac output syndrome (LCOS) is a common complication in cardiac surgery after weaning from cardiopulmonary bypass (CPB) associated with high morbidity and mortality. Its prompt recognition and management may mitigate the effect of LCOS on the outcome. To date, advanced age, prolonged CPB, urgent surgery and impaired left ventricular function assessed by left ventricular ejection fraction (LVEF) are commonly considered strong predictors of postoperative LCOS. Nevertheless, LVEF has several limitations including image quality, operator experience, limited reproducibility, inter- and intra-observer discrepancy and load/volume dependency. Global Longitudinal Strain (GLS), with automated speckle-tracking echocardiography (STE) may overcome several of the LVEF limitations. In fact, while the LVEF detects changes in left ventricular chamber volume, GLS reflects myocardial longitudinal deformation due to contraction. The rate of myocardial deformation over time (expressed as 1/s) is called GLS Rate. Global Longitudinal Strain, mostly evaluated from transthoracic echocardiography (TTE), has shown lower inter- and intra-observer variability, a better reproducibility and prognostic value compared to LVEF in a generic cardiac population. In addition the results of the GLS with TTE (GLS-TTE) may not be shifted in cardiac surgery due to the effect of the general anesthesia (GA) and positive pressure ventilation. Thus, these factors should be considered when the global longitudinal strain, evaluated from transesophageal echocardiography (GLS-TEE) is used as predictor of early outcome. Amabili et al. have shown that GLS-TEE is better than LVEF in predicting LCOS in a general cardiac surgery population. Similarly Sonny et al. in patients undergoing aortic valve surgery for stenosis have reported that a GLS-TEE and GLS-TEE Rate are superior to standard echocardiographic parameters in predicting a complicated course. To the best of our knowledge, there are no studies investigating the role of intraoperative evaluation of GLS-TEE and GLS-TEE Rate as predictors of LCOS in mitral valve surgery. In this setting LVEF is not a reliable marker of cardiac function due to a systematic overestimation of the ejection fraction. Moreover these patients are at high risk of postoperative cardiac dysfunction and LCOS owing to the afterload mismatch after mitral surgery. For the reasons mentioned above, more effective predictors are advocated. In the present study we try to fill the gap. Thus, aim of present study is to assess the role of GLS-TEE, GLS-TEE Rate and standard echocardiographic parameters in predicting LCOS in on-pump mitral surgery. In doing so, the best cut-off for each echocardiographic parameter will be provided. Finally to detect the effect of the GA, the echocardiographic parameters calculated after the induction of GA will be compared with those collected preoperatively.

A telephonic follow-up will be performed at 30 days and 12-months investigating mortality and rehospitalization due to heart failure.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective or urgent open mitral valve repair or mitral valve replacement over 18 years
* Ability to sign informed consent
* Availability of pre-CBP and after-CPB intraoperative transesophageal echocardiography which include a 4-chambers, 2-chambers and a long axis view at a minimum frame rate of 50 Hz
* Good quality echocardiographic images with a optimal endocardial definition
* Good quality ECG tracing

Exclusion Criteria:

* All patients undergoing emergent open mitral valve repair or mitral valve replacement
* Unavailability of pre-CBP and after-CPB intraoperative transesophageal echocardiography which include a 4-chambers, 2-chambers and a long axis view at a minimum frame rate of 50 Hz
* Poor quality echocardiographic images
* ECG artefacts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open mitral valve repair or mitral valve replacement over 18 years old at Scientific Institute San Raffaele will be asked for their informed consent and enrolled in the present study.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Global longitudinal strain of myocardium in mitral valve surgery | Intraoperative 6 hours
  Offline processing of GLS, GLS Rate
Number of patients with low cardiac output syndrome after mitral valve surgery | 30 days
Global longitudinal strain threshold associated with LCOS after mitral valve surgery | Intraoperative 6 hours

SECONDARY OUTCOMES:
Effect of general anesthesia on systole and diastole | Intraoperative 6 hours
All-cause mortality during the follow-up | 30 days and 1years
Length of intensive care unit stay | 30 days
Length of hospital stay | 30 days
30-day or in hospital mortality | 30 days
Duration of post-operative mechanical ventilation | 30 days
Post-operative rate of acute kidney injury | 30 days
Post-operative rate of hepatic dysfunction | 30 days
Readmission rate in intensive care | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute San Raffaele, Milan, Italy

REFERENCES:
- [Result] Sonny A, Alfirevic A, Sale S, Zimmerman NM, You J, Gillinov AM, Sessler DI, Duncan AE. Reduced Left Ventricular Global Longitudinal Strain Predicts Prolonged Hospitalization: A Cohort Analysis of Patients Having Aortic Valve Replacement Surgery. Anesth Analg. 2018 May;126(5):1484-1493. doi: 10.1213/ANE.0000000000002684. PMID 29200066
- [Result] Amabili P, Benbouchta S, Roediger L, Senard M, Hubert MB, Donneau AF, Brichant JF, Hans GA. Low Cardiac Output Syndrome After Adult Cardiac Surgery: Predictive Value of Peak Systolic Global Longitudinal Strain. Anesth Analg. 2018 May;126(5):1476-1483. doi: 10.1213/ANE.0000000000002605. PMID 29116972
- [Derived] Monaco F, Bonaccorso A, D'Andria Ursoleo J, Pruna A, Lerose CC, Di Prima AL, Barucco G, Landoni G, Licheri M; Mit-Go Study Group Collaborators. Intraoperative global longitudinal strain and strain rate as predictors of unfavorable outcome following on-pump mitral surgery: a prospective observational study. J Anesth Analg Crit Care. 2025 Oct 22;5(1):70. doi: 10.1186/s44158-025-00288-1. PMID 41126360